CLINICAL TRIAL: NCT00510003
Title: A Multicenter, 3-week, Randomized, Double-blind, Parallel-group, Vehicle-controlled Study to Evaluate the Efficacy and Safety of Pimecrolimus Cream 1% in Pediatric Patients With Mild to Moderate Atopic Dermatitis
Brief Title: Assessment of Pruritus Improvement With Pimecrolimus Treatment on the Areas Affected by Mild-to-moderate AD, in Patients 2- to 11- Year-old
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CASM981CES02
Record Dates: First submitted 2007-07-31; First posted 2007-08-01 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis, children, pimecrolimus, eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — pimecrolimus

INTERVENTIONS:
Drug: Pimecrolimus — Pimecrolimus cream 1 %
  Other Names: Elidel

SUMMARY:
The purpose of this study is to assess the efficacy and safety of pimecrolimus cream 1% in relation to the improvement of pruritus in pediatric patients (2- to 11- year-old) with mild to moderate atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Age: between 2 - 12 years.
* Outpatients with diagnosis of atopic dermatitis
* Atopic dermatitis affecting ≥ 5% of Total Body Surface Area at Baseline Investigator's Global Assessment score of 2 (mild) or 3 (moderate).
* Baseline visit pruritus (itching) severity assessment score of 2 (moderate) or 3 (severe).
* Patients or patient's legal guardian who has been informed of the study procedures and has signed the informed consent form approved for the study prior to starting any study related procedures, including washout (in case that it would be necessary).

Exclusion Criteria:

* Patients being breast-fed by women receiving systemic or prohibited medication.
* Children with known hypersensitivity to study medication.
* Children who received phototherapy or systemic therapy (immunosuppressants, cytostatics) known to affect atopic dermatitis within the previous month or topical therapy (tar, topical corticosteroids), systemic corticosteroids, systemic antibiotics or leukotriene antagonists within the previous week.
* Children who received investigational drugs within 8 weeks prior to first application of study medication.
* Children who had concurrent skin disease or active bacterial, viral or fungal infection.
* Immunocompromised children (e.g., lymphoma, AIDS, Wiskott-Aldrich Syndrome) or children with a history of malignant disease.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 2 Years to 12 Years | Sex: All
Age Groups: Child
Enrollment: 117 (Actual)
Dates: Start 2004-12; Primary Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Change in pruritus Visual Analogic Scale (VAS) with respect to the basal score between and within treatment groups, daily evaluation.

SECONDARY OUTCOMES:
• Reduction ≥ 50% in pruritus VAS with respect to basal score (responding patients) between groups and within groups (daily evaluation). • Change in sleep quality VAS in the pimecrolimus group with respect to the basal score (daily evaluation), and

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis Pharma AG, Basel, Switzerland
Locations (1):
- Novartis Investigative Site, Madrid, Spain